CLINICAL TRIAL: NCT04011449
Title: State-dependent Pathophysiological Oscillations in Parkinson's Disease and Treatment With DBS Using the Medtronic RC+S
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUR-2019-27724
Record Dates: First submitted 2019-06-10; First posted 2019-07-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease; Parkinson
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device Implantation (Experimental): Implantation of the Medtronic RC+S Deep Brain Stimulation (DBS) system
  Interventions: Device: Medtronic RC+S DBS system

INTERVENTIONS:
Device: Medtronic RC+S DBS system — Implantation of the Medtronic RC+S Deep Brain Stimulation (DBS) system

SUMMARY:
Primary objectives.

The ability of the RC+S to record Local Field Potentials (LFP's) is novel in Deep Brain Stimulation (DBS) technology. The primary goals of this project are to use this function of the RC+S to characterize:

1. The state- and target-dependency of neuronal oscillations in the subthalamic nucleus (STN), internal globus pallidus (GPi) or external globus pallidus (GPe) of patients with PD,
2. How these oscillations are altered by levodopa,
3. The effects of unilateral standard clinical isochronal (e.g. 140 Hz) GPi-, GPe-, and STN-DBS on oscillatory activity and its relationship to the presence and severity of parkinsonian motor signs.

These experiments will leverage the capacity to record LFPs from macroelectrodes implanted in either the GPi/GPe or STN using the Medtronic RC+S DBS system. The long-term goal for this project is to develop closed-loop methods for DBS that are state (resting vs. movement) and movement-phase appropriate.

Secondary objectives.

In addition to establishing the relationship between neural oscillations in the STN, GPi and GPe to clinical and quantitative measures of akinesia, bradykinesia, tremor and rigidity, this project will also examine the relationship of neural oscillations to:

1. Levodopa-resistant motor features such as postural instability and gait (including freezing of gait),
2. Response inhibition and impulse control.

DETAILED DESCRIPTION:
The Olympus Research System (RC+S) is an implantable pulse generator (IPG) designed to deliver deep brain stimulation (DBS) like a standard clinical neurostimulator, but which allows recordings of local field potential (LFP) activity from the implanted DBS lead.

LFPs are composite electrical signals generated by the brain. They are conventionally divided into frequency bands, as follows: 0-3 Hz (delta), 4-7 Hz (theta), 8-12 Hz (alpha), 13-30 Hz (beta), 31-200 Hz (gamma), and >200 Hz (high frequency). The instantaneous amplitude and power of the LFP recordings are believed to represent the degree of synchronization among neurons surrounding the electrode. A transient increase in power in a particular band, in response to a behavioral event, is called an event-related synchronization (ERS), while a transient decrease in power is called event-related desynchronization (ERD). ERD and ERS are typically calculated by averaging the power across time segments and comparing this average to a reference epoch.

Research staff at the University of Minnesota will follow FDA guidelines for software development for the RC+S.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD.
* Age 45-75 years
* Demonstrated good response (≥ 30%) to Sinemet or dopamine agonist medications as assessed by total UPDRS III score (off and on meds)
* Clinical plan for unilateral STN- or GPi-DBS surgery to treat their clinical motor signs within the next four months
* Written documentation of willingness to participate in the study per protocol as evidenced by the informed consent process

Exclusion Criteria:

* Clinically significant medical disease that would increase the risk of developing pre- or post-operative complications (e.g., major cardiac or pulmonary disease)
* Evidence of secondary or atypical parkinsonism
* Dementia as evidenced by impairment in two neuropsychological domains and impaired or borderline neuropsychological function in one additional domain.
* Unable to undergo MR imaging (e.g., due to incompatible implanted pacemaker)
* Previous pallidotomy or DBS surgery
* Women who are currently pregnant
* MRI brain abnormalities that could indicate a neurological disorder other than idiopathic Lewy body Parkinson's disease.
* Subjects with severe or poorly controlled depression defined according to DSM-V criteria and a scored on a validated depression assessment scale.
* Epilepsy
* Immunocompromised
* Requires diathermy, electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) to treat a chronic condition
* Has an implanted electronic device such as a neurostimulator, cardiac pacemaker or medication pump.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Passive and Active Rigidity Quantification | 6-months
  Peak resistive torque integral of resistive torque over the pronation and supination Range of Motion (ROM)
Ballistic Elbow Flexion to a Target: Peak Velocity | 6-months
  Peak velocity
Ballistic Elbow Flexion to a Target: Stop Reaction Time | 6-months
  Stop reaction time
Rapid Alternating Pronation-Supination Movements: RMS | 6-months
  Root Mean Square (RMS)-Displacement RMS
Rapid Alternating Pronation-Supination Movements: Freezing Episodes Duration | 6-months
  Duration of hesitation or arrest (freezing) episodes
Rapid Alternating Pronation-Supination Movements: Freezing Episodes Number | 6-months
  Number of hesitation or arrest (freezing) episodes
Gait: Step length | 6-months
  Step length
Gait: Step Time | 6-months
  Step time
Gait: Double Support Time | 6-months
  Double support time
Gait: Obstacles | 6-months
  Percentage of obstacles successfully avoided
Gait: Freezing Episodes Duration | 6-months
  Duration of freezing episodes
Gait: Freezing Episodes Number | 6-months
  Number of freezing episodes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No